CLINICAL TRIAL: NCT04605770
Title: A Single-Arm, Multicenter, Open-Label, Phase 2 Study of Pemetrexed/Cisplatin Chemotherapy for Patients With Metastatic/Recurrent Soft Tissue Sarcoma in 4- Independent Histologic Subtypes
Brief Title: Pemetrexed, Cisplatin With Soft Tissue Sarcoma
Acronym: ALBATROSS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyo Song Kim, Principal investigator, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0923
Record Dates: First submitted 2020-10-19; First posted 2020-10-28 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pemetrexed+cisplatin (Experimental): Pemetrexed 500 mg/m2 (Day 1) and cisplatin 75 mg/m2 (Day 1) will be given via intravenous (IV) infusion. Each cycle consists of 21 days, and this combination therapy will be continued until Cycle 6. Starting from Cycle 7, pemetrexed alone will be administered every 3 weeks (Q3W) as IV infusion until disease progression.
  Interventions: Drug: pemetrexed+cisplatin

INTERVENTIONS:
Drug: pemetrexed+cisplatin — Pemetrexed 500 mg/m2 (Day 1) and cisplatin 75 mg/m2 (Day 1) will be given via intravenous (IV) infusion. Each cycle consists of 21 days, and this combination therapy will be continued until Cycle 6. Starting from Cycle 7, pemetrexed alone will be administered every 3 weeks (Q3W) as IV infusion until disease progression.
  Vitamin B12 1000 mcg intramuscular (IM) injection will be given within 14 days prior to the first dose of pemetrexed, every 9 weeks (on the same day as study treatment) thereafter, and then 21 days after the last dose of pemetrexed. Folic acid 1 mg will be administered daily starting from 14 days before the first dose of pemetrexed and continued until 21 days after the last dose of pemetrexed. Study treatment will be continued until PD, unacceptable AE, or decision to discontinue by subject or physician.

SUMMARY:
Soft tissue sarcoma (STS) is rare malignancy of mesodermal origin, representing less than 1% of all malignant neoplasms. They are a group of diseases encompassing diverse histological subtypes with very different biomorphologies, prognoses, and responses to treatments. At advanced stages of STS, anticancer treatments are less effective and the prognosis is poor with a median survival of 8 to 18 months. Doxorubicin and ifosfamide given each alone or in their combination have represented the mainstream of anticancer treatments in metastatic STS. However, salvage treatments for patients with progression after doxorubicin/ifosfamide-based treatment are limited and anticancer agents such as gemcitabine/docetaxel, pazopanib, eribulin and trabectedin are currently used as a standard of care (SOC).

For metastatic sarcoma, a study of pemetrexed alone in patients with refractory STS who have progressed after doxorubicin and/or ifosfamide-based anticancer treatment was conducted. In this study including 48 patients, most of whom had relatively poor course of disease with disease progression after the 2nd- and/or 3rd-line treatment, pemetrexed was well tolerated and associated with 5% of response rate and 33% of 3-month progression-free rates suggesting potential antitumor efficacy with good tolerability profile with refractory STS.

However, as conventional agents have showed different efficacy depending on various subtypes of STS, a confirmatory study to see clinical utilities of a given regimen by subtype is required also for pemetrexed/cisplatin. Therefore, the investigators intend to proceed this phase 2 clinical trial to evaluate the efficacy and safety of pemetrexed/cisplatin combination therapy in patients with advanced/metastatic STS who received up to two-lines of prior palliative anticancer treatments with histological subtype-specific cohorts (leiomyosarcoma, synovial sarcoma, malignant peripheral nerve sheath tumor, and others) in order to provide a basis for a subsequent phase 3 study by selecting histological subtype(s) in which the efficacy of study regimen is to be proven.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed, advanced/metastatic STS
* Is ≥ 19 years of age
* Eastern Cooperative Oncology Group performance status of 0 or 1
* measurable disease per Response Evaluation Criteria in Solid Tumors Version 1.1
* laboratory values indicating adequate organ function
* a documented postmenopausal woman, or is a premenopausal woman with negative urine or serum pregnancy test
* life expectancy ≥ 12 weeks

Exclusion Criteria:

* previously received more than 2 regimens of cytotoxic chemotherapy
* received chemotherapy, surgery to major organ, or radiotherapy within the last 2 weeks
* ongoing toxicity (≥ CTCAE grade 2) from previous anticancer therapy
* central nervous system (CNS) metastases requiring active treatment
* diagnosis of second malignancy or has a history of active malignancy within the past 3 years
* other medical conditions where the study treatment is intolerable
* history of active infection
* hypersensitivity to pemetrexed or any of its excipients
* Co-administration with yellow fever vaccine
* pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate | at 12 weeks
  Progression-free survival rate at Week 12 (PFR 12) based on RECIST 1.1

SECONDARY OUTCOMES:
overall response rate | every 6 weeks, up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea